CLINICAL TRIAL: NCT02515084
Title: Preliminary Study of the Interest of Diffusion-weighted Magnetic Resonance Imaging in the Early Detection of Differentiated Thyroid Carcinoma Cervical Recurrence. Comparison with18F-FDG PET/CT
Brief Title: Comparison DW-MRI vs FDG PET/CT in the Detection of Early Recurrence of Cervical Well-differentiated Thyroid Carcinoma
Acronym: THYRIRMTEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHB 10-03
Record Dates: First submitted 2015-07-24; First posted 2015-08-04 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Thyroid Cancer; Relapse
Keywords: recurrence Thyroid cancer; 18F-FDG PET-CT; diffusion-weighted Magnetic Resonance Imaging
MeSH Terms: conditions — Thyroid Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FDG-PET and dw-MRI (Experimental): At the inclusion, both all patients, a 18F-FDG-PET/CT and a dw-MRI will be performed
  Interventions: Device: PET; Device: MRI imaging

INTERVENTIONS:
Device: PET — A FDG PET scan and a diffusion-weighted Magnetic Resonance Imaging will be performed to compare the efficacy to diagnose relapse in thyroid carcinoma
Device: MRI imaging

SUMMARY:
The purpose of the study is to evaluate the concordance between the 18F-PET/CT under thyrotropin stimulation and the diffusion-weighted Magnetic Resonance Imaging, in the detection of residual mass in 40 patients with partial response or relapsed differentiated thyroid carcinoma.

DETAILED DESCRIPTION:
The schedule and the procedures of the study are the following ones :

* Baseline evaluation :

  * Clinical examination with neck echography after rhTSH stimulation
  * Normal whole body scan
* First visit (inclusion):

  18F-FDG PET/CT DW-MRI of the neck if possible performed shortly after the PET CT or within following days
* Following visits: at 6 months and 12 months

  * DW-MRI of the neck performed shortly after the PET CT or within following days.
  * Ultrasonography guided fine needle aspiration for cytology for detection of cervical metastases and identifying thyroglobuline in the needle washout fluid if needed and in case of positivity of either PET or DW-MRI exams.
  * Histological assessment of biopsies if performed

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Subjects must be 18 years of age or older,
* Histologically confirmed papillary or follicular differentiated thyroid carcinoma with partial response or complete response, defined by

  * Thyroglobulin > 2 μg/L under thyrotrophin stimulation, four months after at least two 131-I based treatments (3,7 GBq/100mCi or more if optimal conditions),
  * Negative extension assessment (total body bone scan, (3,7 GBq/100 mCi or more)), echography, CT scan ( neck, thorax, abdomen): no findings..
* Patient's Informed Consent form signed.

Exclusion Criteria:

* History of previous cancer within the least three years,
* Performance Status > 2,
* Protected adults
* Any medical, psychological, social or disabling conditions that could interfere or jeopardize the patient's participation
* History of allergy to radio-iodine,
* Estimated GFR < 45 ml/min /m² (MDRD method),
* Women of childbearing potential without contraceptive method,
* Uncontrolled diabetes mellitus,
* Hypersensitivity to FDG or to any radio-tracers,
* Contraindication to administration of Thyrogen® 0.9mg
* Intraocular foreign bodies or any metallic foreign bodies that contraindicates the MRI.
* Vascular clips, any object or implanted device that could interact with the ferromagnetic field,
* Coronary and peripheral clips, aortic stent grafts, prosthetic heart valves, annuloplasty rings, vena cava filters, cardiac pacemaker, implantable cardiovascular defibrillators....,
* Implanted insulin infuser
* Neurostimulator device
* Claustrophobia
* Agitation or psychological trouble

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Report of positive or negative results of detection of recurrent lesions from both dw-MRI and 18F-FDG PET/CT. data will be reported extensively and descriptively. | 1 year
  To assess concordance between FDG PET-CT scan and MRI in detection of cervical residual masses in 40 patients in Partial Response or in relapse cervical well-differentiated thyroid carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Vera, MD, PhD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France